CLINICAL TRIAL: NCT02788188
Title: A Phase 1, Randomized Double-Blind, Placebo-Controlled, Single Ascending Dose Safety, Tolerability, and Pharmacokinetics Study of SAB-301 in Healthy Adults
Brief Title: Safety, Tolerability, and Pharmacokinetics of SAB-301 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Naval Medical Research Center (U.S. Federal Agency); SAb Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 160119; 16-I-0119
Record Dates: First submitted 2016-05-28; First posted 2016-06-02 (Estimated); Results first posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2017-07

CONDITIONS: Middle East Respiratory Syndrome Coronavirus
Keywords: First in Human; Middle East Respiratory Syndrome (MERS); Tc Bovine-Derived; Transchromosomic Cattle
MeSH Terms: conditions — Coronavirus Infections | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1 (Experimental): Cohort 1: 1mg/kg SAB-301 in normal (9%) saline; concentration 1mg/mL (0.1%)
  Interventions: Biological: SAB-301
- Placebo (Placebo Comparator): Normal (0.9%) saline in approximately the same volume as each cohort in the experimental drug arm.
  Interventions: Other: Normal (9%) Saline
- Cohort 2 (Experimental): Cohort 2: 2.5 mg/kg SAB-301 in normal (9%) saline; concentration 1mg/mL (0.1%)
  Interventions: Biological: SAB-301
- Cohort 3 (Experimental): Cohort 3: 5mg/kg SAB-301 in normal (9%) saline; concentration 4mg/mL (0.4%)
  Interventions: Biological: SAB-301
- Cohort 4 (Experimental): Cohort 4: 10mg/kg SAB-301 in normal (9%) saline; concentration 4mg/mL (0.4%)
  Interventions: Biological: SAB-301
- Cohort 5 (Experimental): Cohort 5: 20mg/kg SAB-301 in normal (9%) saline; concentration 20mg/mL (2%)
  Interventions: Biological: SAB-301
- Cohort 6 (Experimental): Cohort 6: 50mg/kg SAB-301 in normal (9%) saline; concentration 20mg/mL (2%)
  Interventions: Biological: SAB-301

INTERVENTIONS:
Biological: SAB-301 — SAB-301 is a purified human immune globulin G (hIgG) polyclonal antibody designed to specifically bind to the MERS-CoV spike (S) protein, a component of the virion membrane that is responsible for binding of the virus to the host cell. The hIgG is purified from the plasma of immunized transchromosomic (Tc) bovines that were immunized with a recombinant spike protein produced in insect cells. SAB-301 is purified hIgG in a sterile liquid formulated in 10 mM glutamic acid monosodium salt, 262 mM D-sorbitol, 0.05 mg/mL Tween 80, pH 5.5. The drug product will be administered intravenously and will be diluted in saline per the clinical protocol.
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4; Cohort 5; Cohort 6
Other: Normal (9%) Saline — Normal (0.9%) saline in approximately the same volume as each cohort in the experimental drug arm.
  Arms: Placebo

SUMMARY:
Background:

Middle East Respiratory Syndrome (MERS) is a newly discovered contagious and sometimes fatal respiratory virus. People often get MERS through close contact with an infected person. Scientists are worried that MERS may spread and cause more infections. There are no vaccines or treatments for MERS right now. Researchers think a new therapy called SAB-301 may be able to help. Antibodies are proteins the body makes to attack viruses. SAB-301 is made of antibodies made in cows to fight MERS. The antibodies are collected from plasma, the liquid part of cow blood.

Objective:

To evaluate the safety and tolerability of SAB-301 in healthy adults.

Eligibility:

Healthy people ages 18 60 who:

Do not have chronic medical problems

Do not take any medications (exceptions are acetaminophen, ibuprofen, vitamins, seasonal allergy meds and oral contraception)

Do not have allergies to beef products

Agree to use two forms of contraception while on study (both men and women)

Design:

Participants will be screened with:

Medical history

Physical examination

Blood and urine tests

Participants will have a return visit.

They will have a physical exam and blood tests.

They will be randomly assigned to receive either SAB-301 or a placebo which is given by infusion

through an arm vein over 1 3 hours.

They will be monitored at the clinic for 6 hours after the infusion. They will have additional blood draws.

Participants will have 2-hour visits 1, 3, 7, 21, 42, and 90 days after the infusion. At each visit they will be evaluated and have blood and urine tests.

DETAILED DESCRIPTION:
The administration of convalescent plasma or hyperimmune immunoglobulin is often used for treatment of emerging infectious diseases. However, production of large quantities of anti-pathogen human plasma and/or immunoglobulin with high affinity and avidity antibodies currently requires donations by convalescent humans, a process that can limit availability for a number of reasons. One novel alternative source is transchromosomic (Tc) cattle that produce fully human polyclonal IgG (hIgG) de novo and mount a robust antibody immune response after vaccination.

This study will evaluate the safety, tolerability, and immunogenicity of SAB-301, a fully human polyclonal anti-MERS IgG collected from transchromosomic cattle. Beginning with a low single-dose, subjects are randomized to receive either SAB-301 or a normal saline control, and evaluated on Study Days 1, 3, 7, 21, 42, and 90. The safety and tolerability is evaluated using symptoms, clinical laboratory tests, pharmacokinetics, and immunogenicity assays. Utilizing a series of stopping rules and a medical monitor, the dose will be escalated as safety and tolerability are established.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age greater than or equal to 18 years and less than or equal to 60 years
  2. Body mass index (BMI) of 19-32 kg/m(2)
  3. Estimated glomerular filtration rate greater than or equal to 70 mL/min at screening, calculated using the CKD-EPI formula
  4. Subjects must agree to:
* Not take any prescription or OTC medications with the exception of acetaminophen, ibuprofen, vitamins, seasonal allergy medications, and/or contraceptive medications for a period 7 days prior to study drug administration (i.e., Day 0)

  5. One of the following in order to avoid pregnancy:
* Females who are able to become pregnant (i.e., are not postmenopausal, have not undergone surgical sterilization, and are sexually active with men) must agree to use at least 2 effective forms of contraception from the date of the subject s signing of the informed consent form through 60 days after the last dose of study drug. At least one of the methods of contraception should be a barrier method.
* Males who have not undergone surgical sterilization and are sexually active with women must agree to use condoms plus have a partner use at least one additional effective form of contraception from the date of the subject s signing of the informed consent form through 60 days after the last dose of study drug.

EXCLUSION CRITERIA:

1. Any history of allergy, anaphylaxis, or severe reaction to beef products (including milk and gelatin)
2. Any history of allergy, anaphylaxis, or severe reaction to IGIV or human blood products
3. Any chronic medical problem that requires daily oral medications (except Tylenol, ibuprofen, oral contraceptives, vitamins, and seasonal allergy medications).
4. History of cardiovascular disease, cardiomyopathy, heart failure, or unexplained syncope
5. Subjects that have had confirmed MERS
6. Women who are breast-feeding
7. Positive urine or serum pregnancy test
8. Abnormal chemistry panel

   -defined as any clinically significant baseline Grade 1 or greater toxicity, or any Grade 3 or greater toxicity (regardless of clinical significance) by the toxicity table

   --evaluating only sodium (Na), potassium (K), serum bicarbonate (total CO2), blood urea nitrogen (BUN), creatinine, glucose, asp (ALT), aspartate aminotransferase (AST), total bilirubin, lactate dehydrogenase (LDH), and estimated glomerular filtration rate (GFR) by the CKD-EPI equation.
9. Abnormal complete blood count (CBC)

   -defined as any clinically significant baseline Grade 1 or greater toxicity, or any Grade 3 or greater toxicity (regardless of clinical significance) by the toxicity table--evaluating only the WBC (to include absolute neutrophil, lymphocyte, and eosinophil counts), hemoglobin, hematocrit, and platelets.
10. Abnormal urinalysis

    -defined as any clinically significant baseline Grade 1 or greater toxicity--evaluating only protein, and RBCs
11. Positive rheumatoid factor
12. IgA deficiency (defined as IgA < 7 mg/dL)
13. Participation in another research study with receipt of any investigational drug within 5 half-lives or 30 days, whichever is longer, prior to study drug administration (i.e., Day 0) and until completion of the study
14. Participation in any other research study for 30 days after study drug administration
15. Receipt of blood products within 2 months prior to study drug administration (i.e. Day 0)
16. Receipt of any vaccination within 30 days prior to study drug administration (i.e. Day 0)
17. Any acute or chronic condition that, in the opinion of the Investigator, would limit the subject s ability to complete and/or participate in this clinical study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2016-05-28; Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Davey, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Luke T, Wu H, Zhao J, Channappanavar R, Coleman CM, Jiao JA, Matsushita H, Liu Y, Postnikova EN, Ork BL, Glenn G, Flyer D, Defang G, Raviprakash K, Kochel T, Wang J, Nie W, Smith G, Hensley LE, Olinger GG, Kuhn JH, Holbrook MR, Johnson RF, Perlman S, Sullivan E, Frieman MB. Human polyclonal immunoglobulin G from transchromosomic bovines inhibits MERS-CoV in vivo. Sci Transl Med. 2016 Feb 17;8(326):326ra21. doi: 10.1126/scitranslmed.aaf1061. PMID 26888429
- [Background] Steinberger BA, Ford SM, Coleman TA. Intravenous immunoglobulin therapy results in post-infusional hyperproteinemia, increased serum viscosity, and pseudohyponatremia. Am J Hematol. 2003 Jun;73(2):97-100. doi: 10.1002/ajh.10325. PMID 12749010
- [Result] Beigel JH, Voell J, Kumar P, Raviprakash K, Wu H, Jiao JA, Sullivan E, Luke T, Davey RT Jr. Safety and tolerability of a novel, polyclonal human anti-MERS coronavirus antibody produced from transchromosomic cattle: a phase 1 randomised, double-blind, single-dose-escalation study. Lancet Infect Dis. 2018 Apr;18(4):410-418. doi: 10.1016/S1473-3099(18)30002-1. Epub 2018 Jan 9. PMID 29329957
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-I-0119.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: 1.0mg/kg: SAB-301 1 mg/kg IV single infusion
- Cohort 2: 2.5mg/kg: SAB-301 2.5 mg/kg IV single infusion
- Cohort 3: 5mg/kg: SAB-301 5 mg/kg IV single infusion
- Cohort 4: 10mg/kg: SAB-301 10 mg/kg IV single infusion
- Cohort 5: 20mg/kg: SAB-301 20 mg/kg IV single infusion
- Cohort 6: 50mg/kg: SAB-301 50 mg/kg IV single infusion
- Placebo: Normal Saline IV single infusion
Period: Overall Study
Arm/Group | Cohort 1: 1.0mg/kg | Cohort 2: 2.5mg/kg | Cohort 3: 5mg/kg | Cohort 4: 10mg/kg | Cohort 5: 20mg/kg | Cohort 6: 50mg/kg | Placebo
Started | 2 | 2 | 4 | 4 | 8 | 8 | 10
Completed | 2 | 2 | 4 | 4 | 8 | 8 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: 1.0mg/kg | Cohort 2: 2.5mg/kg | Cohort 3: 5mg/kg | Cohort 4: 10mg/kg | Cohort 5: 20mg/kg | Cohort 6: 50mg/kg | Placebo | Total
Number analyzed (Participants) | 2 | 2 | 4 | 4 | 8 | 8 | 10 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4 | 4 | 8 | 8 | 10 | 38
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 3 | 3 | 4 | 3 | 3 | 18
  Male | 2 | 0 | 1 | 1 | 4 | 5 | 7 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 3
  Not Hispanic or Latino | 2 | 2 | 4 | 3 | 7 | 7 | 10 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 0 | 2 | 0 | 2 | 6
  White | 2 | 2 | 2 | 4 | 5 | 7 | 4 | 26
  More than one race | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Having Adverse Events
Description: Number of participants who experienced an adverse event
Time Frame: 90 days
Population: Number of participants who completed both treatment and placebo
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: 1.0mg/kg | Cohort 2: 2.5mg/kg | Cohort 3: 5mg/kg | Cohort 4: 10mg/kg | Cohort 5: 20mg/kg | Cohort 6: 50mg/kg | Placebo
Number analyzed (Participants) | 2 | 2 | 4 | 4 | 8 | 8 | 10
Participants | 1 | 2 | 2 | 4 | 7 | 8 | 10

ADVERSE EVENTS:
Time Frame: 90 Days
Arm/Group | Cohort 1: 1.0mg/kg | Cohort 2: 2.5mg/kg | Cohort 3: 5mg/kg | Cohort 4: 10mg/kg | Cohort 5: 20mg/kg | Cohort 6: 50mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/4 | 0/4 | 0/8 | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/4 | 0/4 | 0/8 | 1/8 | 0/10
Other Adverse Events (participants affected / at risk) | 1/2 | 2/2 | 2/4 | 4/4 | 7/8 | 8/8 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: 1.0mg/kg (N=2) | Cohort 2: 2.5mg/kg (N=2) | Cohort 3: 5mg/kg (N=4) | Cohort 4: 10mg/kg (N=4) | Cohort 5: 20mg/kg (N=8) | Cohort 6: 50mg/kg (N=8) | Placebo (N=10)
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: 1.0mg/kg (N=2) | Cohort 2: 2.5mg/kg (N=2) | Cohort 3: 5mg/kg (N=4) | Cohort 4: 10mg/kg (N=4) | Cohort 5: 20mg/kg (N=8) | Cohort 6: 50mg/kg (N=8) | Placebo (N=10)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chlamydial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1 | 2
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin candida (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tinea capitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood bicarbonate decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1 | 1
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 3
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood sodium decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 1 | 2 | 1 | 1 | 2
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Albuminuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 2 | 2 | 2
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT02788188/Prot_SAP_000.pdf